CLINICAL TRIAL: NCT02756858
Title: An Extension Study of ANAVEX2-73 in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANAVEX2-73-003
Record Dates: First submitted 2016-03-08; First posted 2016-04-29 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tetrahydro-N, N-dimethyl-2,2-diphenyl-3-furanmethanamine hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ANAVEX2-73 Oral as assigned in ANAVEX2-73-002 (Experimental)
  Interventions: Drug: ANAVEX2-73

INTERVENTIONS:
Drug: ANAVEX2-73

SUMMARY:
This open label extension study is designed to provide continued access to ANAVEX 2-73 for eligible subjects with mild to moderate Alzheimer's Disease who have previously participated in the Anavex sponsored study ANAVEX2-73-002.

ELIGIBILITY:
Inclusion Criteria:

* Previous exposure to ANAVEX2-73 via participation in Phase 2a Study of ANAVEX2-73 Adaptive-Trial-Design With Repeated Doses, MTD Finding, Pharmacodynamic and Bioavailability Evaluation in Patients With Mild to Moderate Alzheimer's Disease With a 12-Month Open Label Follow-Up Period (ANAVEX2-73-002)

Exclusion Criteria:

* Have not previously participated Phase 2a Study of ANAVEX2-73 Adaptive-Trial-Design With Repeated Doses, MTD Finding, Pharmacodynamic and Bioavailability Evaluation in Patients With Mild to Moderate Alzheimer's Disease With a 12-Month Open Label Follow-Up Period (ANAVEX2-73-002)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-03; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 208 weeks
  Safety

SECONDARY OUTCOMES:
Score from MMSE (Mini-mental state examination score) | Baseline; Weeks: 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156, 169, 182, 195, 208
  Exploratory Efficacy
Score from ADCS-ADL (Alzheimer's Disease Co-operative Study - Activities of Daily Living Inventory) | Baseline; Weeks: 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156, 169, 182, 195, 208
  Exploratory Efficacy
HAM-D Score (Hamilton Psychiatric Rating Scale for Depression) | Baseline; Weeks: 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156, 169, 182, 195, 208
  Exploratory Efficacy

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Melbourne Health - The Royal Melbourne Hospital, Melbourne, Victoria
  - Austin Health - Heidelberg Repatriation Hospital, Melbourne, Victoria
  - Caulfield Hospital, Melbourne, Victoria
  - Nucleus Network- Centre for Clinical Studies, Melbourne, Victoria
  - St. Vincent's Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Study results will be presented at a scientific conference and/or published.

REFERENCES:
- [Derived] Hampel H, Williams C, Etcheto A, Goodsaid F, Parmentier F, Sallantin J, Kaufmann WE, Missling CU, Afshar M. A precision medicine framework using artificial intelligence for the identification and confirmation of genomic biomarkers of response to an Alzheimer's disease therapy: Analysis of the blarcamesine (ANAVEX2-73) Phase 2a clinical study. Alzheimers Dement (N Y). 2020 Apr 19;6(1):e12013. doi: 10.1002/trc2.12013. eCollection 2020. PMID 32318621